CLINICAL TRIAL: NCT02619032
Title: Remifentanil vs Fentanyl During Day Case Dental Surgery in Persons With Special Needs: a Comparative Study of Their Effect on Stress Response and Postoperative Pain
Brief Title: Remifentanil and Fentanyl in Dental Surgery (REFEDS)
Acronym: REFEDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: Asklepieion Voulas General Hospital (Other Government)
Responsible Party: Principal Investigator, Paraskevi Matsota, Assoc. Prof. of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ATT968
Record Dates: First submitted 2015-11-25; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Pain
Keywords: remifentanil; fentanyl; dental surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Remifentanil; Fentanyl

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Active Comparator): Drug: Remifentanil (Ultiva). Intraoperative intravenous infusion of remifentanil 0.5-1 μg/kg/min for up to 1 h.
  Interventions: Drug: Remifentanil; Drug: Fentanyl
- Fentanyl (Active Comparator): Drug: Fentanyl (FNT). Intraoperative administration of fentanyl given as one single bolus dose of 50 μg at the time of induction of anesthesia.
  Interventions: Drug: Remifentanil; Drug: Fentanyl

INTERVENTIONS:
Drug: Remifentanil — Intraoperative continuous infusion of remifenatanil. Remifentanil infusion was interrupted upon completion of surgical intervention.
  Other Names: Ultiva
Drug: Fentanyl — Fentanyl 50 μg iv bolus at the induction of anesthesia and before the start of surgery.
  Other Names: FNT

SUMMARY:
This study was a prospective comparative study. The purpose of this study was to investigate the hypothesis whether remifentanil compared to fentanyl can induce less inflammatory and stress response to the day-case dental surgery in Persons with special needs (PSN). Secondary aims were to investigate comparatively their effect on patients intraoperative hemodynamic response and postoperative analgesia.

DETAILED DESCRIPTION:
The study included 46 adult patients with cognitive impairment who underwent day-case dental surgery under general anesthesia with propofol aiming to keep a BIS-values range between 40-45. Nasal tracheal intubation was performed in all patients while neuromuscular blockade was achieved by rocuronium 0.6 mg/kg iv and repetitive doses of rocuronium of 10 mg iv, if needed.

Patients were randomly allocated receive for intraoperative analgesia either fentanyl 50 μg iv bolus (group F, n=23) or continuous infusion of remifentanil 0.5-1 μg/kg/min (group R, n=23). Randomization was performed using using a computer-generated randomization schedule.

Intraoperatively, patients in both groups received IV granisetron 3 mg, methylprednisolone 125 mg and clindamycin 600 mg, while atropine 0.02 mg/kg and neostigmine (0.05 mg/kg) was administered to to reverse neuromuscular blockade. Intraoperative monitoring included non-invasive measurement of arterial blood pressure, electrocardiogram, pulse oxymetry, capnography and Bispectral Sedation Index (BIS®).

Postoperatively, patients remained under surveillance in the post-anesthesia care unit [PACU] for 3 h. Postoperative pain was assessed for the first 12 postoperative hours, at 30 min time-intervals for the first 3 hours, and every 3 hours thereafter by an independent observer, blinded to the study group, using the Wong-Baker faces pain rating scale (0-6). If pain scores were ≥3 a rescue dose of paracetamol 12.5 mg/kg iv was administered.

Inflammation markers and stress hormones [cortisol, Tumor necrosis factor (TNF-a), substance-P, melatonin and β-endorphin] were measured in each patient before induction of anesthesia, after tracheal intubation and at the end of operation.

Statistical Analysis was performed using Kolmogorov-Smirnov test, Student's unpaired t-test or Repeated Measures ANOVA with Holm's post-hoc analysis appropriately. A p value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cognitive impairment
* of category II according to the American Society of Anesthesiology (ASA) classification
* scheduled for elective dental surgery with short duration

Exclusion Criteria:

* Patients of more than category II of American Society of Anesthesiology (ASA) classification
* Prolonged duration of surgery (>1 hour)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2005-10; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline plasma cortisol values at 1 hour | At 1 hour after the induction of anesthesia and surgery
  Plasma cortisol values were measured with an ELISA kit as mg/dl
Change from baseline plasma tumor necrosis factor-α (TNF-α) values at 1 hour | At 1 hour after the induction of anesthesia and surgery
  Tumor necrosis factor-α (TNF-α) measurement was performed with Elisa immunoenzyme assay as pg/ml
Change from baseline plasma substance-P values at 1 hour | At 1 hour after the induction of anesthesia and surgery
  Substance-P measurement was performed with Elisa immunoenzyme assay as ng/ml
Change from baseline plasma melatonin values at 1 hour | At 1 hour after the induction of anesthesia and surgery
  Melatonin measurement was performed with Elisa immunoenzyme assay as pg/ml
Change from baseline plasma β-endorphin values at 1 hour | At 1 hour after the induction of anesthesia and surgery
  β-endorphin was measured with Elisa immunoenzyme assay as ng/ml

SECONDARY OUTCOMES:
Differences in intraoperative systolic arterial blood pressure values (mm Hg) between the two study groups | 1 hour
  Measurements before the induction of anesthesia (baseline values) and at and 60 min (1 hour) after the induction of anesthesia
Differences in intraoperative heart rate values (bmp) between the two study groups | 1 hour
  Measurements before the induction of anesthesia (baseline values) and at 60 min (1 hour) after the induction of anesthesia
Differences in postoperative pain scores scores between the two study groups | Up to 12 postoperative hours
  Pain was assessed using the Wong-Baker faces pain rating scale (0-6) at 12 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Eirini A Sklika, Consultant, Principal Investigator — Asklepeion Voulas General Hospital
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece